CLINICAL TRIAL: NCT00947791
Title: Intravenous Ketamine in Treatment-Resistant Bipolar Depression
Brief Title: Treatment Study of Bipolar Depression
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Change in available resources for study procedures
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, James Murrough, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 08-1422
Record Dates: First submitted 2009-07-27; First posted 2009-07-28 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Depression; Treatment-Resistant; ketamine; antidepressant; glutamate
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Patient, doctor and rater are masked (triple masked). Only the research pharmacist is unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ketamine/Midazolam (Experimental): Patients receive both treatment conditions (ketamine and midazolam) in a single arm, crossover design. Patients are randomized to ketamine-midazolam. Each treatment occurs as a single intravenous infusion on one treatment day. The two treatment conditions occur 2 weeks apart.
  Interventions: Drug: ketamine; Drug: midazolam
- Midazolam/Ketamine (Experimental): Patients receive both treatment conditions (ketamine and midazolam) in a single arm, crossover design. Patients are randomized to midazolam-ketamine. Each treatment occurs as a single intravenous infusion on one treatment day. The two treatment conditions occur 2 weeks apart.
  Interventions: Drug: ketamine; Drug: midazolam

INTERVENTIONS:
Drug: ketamine — a single IV infusion of ketamine, IV 0.5 mg/kg
Drug: midazolam — a single IV infusion of midazolam, 0.045 mg/kg

SUMMARY:
The purpose of this study is to determine whether a single intravenous administration of an N-methyl-D-aspartate antagonist is safe and effective for the acute treatment of bipolar depression.

DETAILED DESCRIPTION:
Bipolar disorder (BPD) is a common, recurrent, and disabling medical condition. Although mania is the defining feature of BPD, depression represents the majority of illness burden in patients with this devastating condition. Despite the high degree of morbidity and mortality associated with bipolar depression, currently available treatments are few and often inadequate. Recently, a single intravenous (IV) dose of the N-methyl-D-aspartate (NMDA) glutamate receptor antagonist ketamine has demonstrated rapid antidepressant effects in severe unipolar depression. Therefore, the objective of the current study is to investigate the safety and efficacy of a single IV dose of ketamine in treatment-resistant bipolar depression (TRBD).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, 21-70 years;
2. Primary diagnosis of bipolar I or II disorder as assessed by the SCID-P and confirmed by a study psychiatrist;
3. Current depressive episode ≥ 8 weeks duration;
4. History of a failure to respond to at least three (3) adequate pharmacotherapy trials in the current depressive episode (see above for definition for adequate trials);
5. Subjects must be on a stable dose of divalproex ER with serum levels greater than 55 mcg/ml prior to enrollment;
6. Subjects must be free of psychotropic medication for at least 2 weeks (4 weeks for fluoxetine) prior to enrollment (with the exception of divalproex ER as above);
7. Subjects must have scored ≥ 32 on the IDS-C30 at both Screening and Infusion Day #1 and #2;

Exclusion Criteria:

1. Women who plan to become pregnant, are pregnant or are breast-feeding;
2. Any unstable medical illness including hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, neurologic, immunologic, or hematologic disease;
3. Clinically significant abnormal findings of laboratory parameters, physical examination, or ECG;
4. Lifetime history of schizophrenia, schizoaffective disorder, OCD, mental retardation, pervasive developmental disorders, or Tourette's syndrome;
5. Current presence of psychotic, mixed or manic symptoms;
6. Lifetime history of antidepressant-induced switch to a manic episode;
7. History of rapid cycling bipolar subtype;
8. Drug or alcohol abuse within the preceding 3 months or dependence within the preceding 5 years;
9. Lifetime exposure to ketamine or phencyclidine;
10. Patients judged by study investigator to be at high risk for suicide.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James W Murrough, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketamine/Midazolam: Participants in this group/condition receive a single IV infusion of ketamine, IV 0.5 mg/kg then 2 weeks later receive Midazolam IV 0.45 mg/kg
- Midazolam/Ketamine: Participants in this group/condition receive a single IV infusion of midazolam, 0.45 mg/kg and then 2 weeks later received single IV infusion of Ketamine 0.50 mg/kg
Period: Overall Study
Arm/Group | Ketamine/Midazolam | Midazolam/Ketamine
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Based on confidentiality concerns, 0 participants analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine/Midazolam | Midazolam/Ketamine | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous
Sex: Female, Male
  Female |  |  | 0
  Male |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Time Frame: 24 hrs post-infusion compared to baseline
Population: Based on confidentiality concerns, 0 participants analyzed.
Arm/Group | Ketamine/Midazolam | Midazolam/Ketamine
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Quick Inventory of Depressive Symptomatology, Self Report (QIDS-SR)
Time Frame: 24 hrs post-infusion compared to baseline
Population: Based on confidentiality concerns, 0 participants analyzed.
Arm/Group | Ketamine/Midazolam | Midazolam/Ketamine
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Young Mania Rating Scale (YMRS)
Time Frame: 24 hrs post-infusion compared to baseline
Population: Based on confidentiality concerns, 0 participants analyzed.
Arm/Group | Ketamine/Midazolam | Midazolam/Ketamine
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Brief Psychiatric Rating Scale (BPRS)
Time Frame: 4 hrs post-infusion compared to baseline
Population: Based on confidentiality concerns, 0 participants analyzed.
Arm/Group | Ketamine/Midazolam | Midazolam/Ketamine
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Clinician-Administered Dissociative States Scale (CADSS)
Time Frame: 4 hrs post-infusion compared to baseline
Population: Based on confidentiality concerns, 0 participants analyzed.
Arm/Group | Ketamine/Midazolam | Midazolam/Ketamine
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Systematic Assessment for Treatment Emergent Effects (SAFTEE)
Time Frame: 4 hrs post-infusion compared to baseline
Population: Based on confidentiality concerns, 0 participants analyzed.
Arm/Group | Ketamine/Midazolam | Midazolam/Ketamine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Adverse Events information not collected
Arm/Group | Ketamine/Midazolam | Midazolam/Ketamine
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes